CLINICAL TRIAL: NCT03208504
Title: A Multi-center Prospective Open-Label Non-Randomized Clinical Study to Evaluate the Safety and Performance of the Single Branch Nexus™ Aortic Arch Stent Graft System.
Brief Title: The Single Branch NEXUS™ Clinical Study
Acronym: NexusSB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP005
Record Dates: First submitted 2017-06-28; First posted 2017-07-05 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Thoracic Aortic Diseases
Keywords: Thoracic Aortic Disease; Thoracic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, non-randomized, interventional clinical study. All subjects will be treated by implantation of the Single Branch Nexus™ Aortic Arch Stent graft System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All subjects in treatment arm will be implanted with the Single Branch Nexus™ Aortic Arch Stent graft System.
  Interventions: Device: Nexus™ Aortic Arch Stent graft

INTERVENTIONS:
Device: Nexus™ Aortic Arch Stent graft — surgical implantation of Nexus™ Aortic Arch Stent graft

SUMMARY:
A prospective, open-label, non-randomized, interventional clinical study, sponsored by Endospan Ltd. Subjects will be followed-up for five years.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and performance of the Single Branch Nexus™ Aortic Arch Stent Graft System for the endovascular treatment of thoracic aortic pathologies requiring landing in the Aortic Arch (zone 0, zone 1, zone2). The investigational device is the Single Branch Nexus™ Aortic Arch Stent Graft System and its designated Delivery System.

Subject population: ten (10) subjects diagnosed with thoracic aortic disease involving the aortic arch, and who have appropriate anatomy to accommodate the Single Branch Nexus™ delivery system in an endovascular procedure. The study will be conducted in 2 clinical sites in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-90.
2. Thoracic aortic pathology requiring landing in the aortic arch (either: zone 0, zone 1, zone2) e.g. aneurysm, stable chronic type B dissection.
3. In patient with a thoracic aneurysm1: dilatation of the aortic arch larger than 5.5cm in diameter, or symptomatic aneurysm of the aortic arch, or aortic diameter growth rate > 5mm per 6 months
4. American Society of Anesthesiologists (ASA) Classification of III & IV or if not eligible for open-repair surgery (for example previous thoracotomy)
5. Patient is considered clinically and hemodynamically stable based on the discretion of the treating physicians.
6. Patient is considered eligible for an elective surgery
7. Access vessels morphology suitable for endovascular repair in terms of tortuosity, calcification and angulation, documented by CTA, MRA:

   * Femoral/Iliac vessel suitable for 20Fr. introducer
   * Brachial/Axial Artery vessel suitable for 8Fr. Introducer
8. To be eligible to receive the SB-Nexus having the following characteristics, as demonstrated on CTA/MRA:

   Access vessels, iliac/femoral & brachial/axillary compatible with vascular access techniques (femoral cutdown or percutaneous), devices, and /or accessories.
   * Access vessels morphology suitable for endovascular repair in terms of tortuosity, calcification and angulation.
   * Cranial Main Module landing zone (at the braceocephalic artery) ≥ 20mm
   * Caudal Main Module landing zone (at the descending aorta) ≥ 30mm
   * Proximal Ascending Module landing zone (at the ascending aorta) ≥ 30mm
9. Patient understands and is voluntarily willing to participate as evidenced by personally signing the Informed Consent document, and willingness to comply with follow-up schedule

Exclusion Criteria:

1. Female is of childbearing potential
2. Life expectancy of less than 5 years due to comorbidities
3. Any medical condition that, according to the investigator's decision, might expose the patient to increased risk by the investigational device or procedure.
4. Patient with complicated anatomy (type IV Aortic arch, mechanical valve with less than 50mm of Ascending Arch).
5. Acutely ruptured or instable aneurysm or an acute vascular injury due to trauma or infected penetrating ulcers of the aorta.
6. Patients with acute (unstable) dissections or mycotic aneurysms, ulcers or intramural hematoma are to be excluded from the study.
7. Patient with an increased risk for aneurysm rupture during the procedure.
8. Patient whose arterial access site is not anticipated to accommodate the access of the Single Branch Nexus™ Delivery System, due to size, tortuosity or hostile groins (scarring, obesity, or previous failed puncture)
9. Patients with severe atherosclerosis or intraluminal thrombus of the aorta or in the BCT
10. Patient is suffering from unstable angina or NYHA classification III and IV and/or ASA classification V and above.
11. Patient has had a myocardial infarction (MI) or cerebral vascular accident (CVA) within 3 months prior to the planned implantation
12. Patient has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to pre-treatment.
13. Patient with a contraindication to undergo angiography
14. Patient with known sensitivities or allergies to the device materials- Nitinol and polyester
15. Clinical conditions that severely inhibit x-ray visualization of the Aorta. Clinical conditions that severely inhibit x-ray visualization of the Aorta like obesity, or other metal stents in proximity to the designated implantation location that can cause artifacts in the x-ray visualization
16. Connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndromes)
17. Patient has history of bleeding diathesis or coagulopathy that may limit the use of dual antiplatelet or anticoagulant therapy by the decision of the investigator. Medical management of patients undergoing endovascular procedures is required for several different reasons. Patients with Aortic pathologies usually have an increased risk of cardiovascular death, necessitating treatment to reduce the overall risk for cardiovascular events. Treatment is in-line with the medical management of coronary artery disease including anti-platelet therapy and sometimes statins. Anti-platelet therapy is also mandatory to prevent complications such as graft-limb thrombosis and peripheral arterial disease (PAD), which is common in such patients.
18. Patient has an active systemic infection at the time of the procedure documented by pain, fever, drainage, positive culture and/or leukocytosis (WBC > 11,000 mm3).
19. Patients who have the condition that threatens to infect the stent graft. The main factors are: immunodepression at the site of the endovascular procedure, treatment of pseudoaneurysms and mycotic aneurysms, presence of neoplasms and use of corticosteroids.
20. Acute renal failure; chronic renal failure (including dialysis); Creatinine > 2.00 mg/dl or > 182 umol/L
21. Patients already treated with an aortic stent graft
22. Patient who underwent major surgery or interventional procedure in the last three months.
23. Patients placed in an institution by authorities or court according to cf. sec 20 para. 1 sentence 4 no. 3 MPG and sec 28d, para 1, sentence 2.
24. Any other medical, social, or psychological issues that in the opinion of the investigator preclude them from receiving this treatment, or the procedures and evaluations pre- and post- treatment.
25. Active participation in another clinical trial.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint - proportion of patients free from MAEs within 30 days | 30 days post implantation
  Proportion of subjects free from MAEs within 30 days post implantation. MAE is defined as: all-cause mortality, myocardial infarction, renal failure, paraplegia, stroke and bowel ischemia for which a causal relationship with the device cannot be excluded on the basis of the adjudication of the independent Data Monitoring Committee (DMC).
Primary Performance Endpoint -Assessment of the rate of successful disease treatment at 30 days | 30 days post implantation
  Assessment of the rate of successful disease treatment at 30 days post implantation, defined as: Successful delivery and deployment of the device, meaning device was deployed and located in the aortic arch isolating the diseased lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kleine, Study Director — Endospan Ltd.
Locations (1):
- Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No